CLINICAL TRIAL: NCT00006656
Title: A Phase I/II Study of the Safety and Tolerability of DTI-015 in Patients With Recurrent Glioblastoma Multiforme
Brief Title: Carmustine in Treating Patients With Progressive or Recurrent Glioblastoma Multiforme
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Direct Therapeutics (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068207; DTI-9901; UCMC-00042402; NCI-V00-1623
Record Dates: First submitted 2000-12-06; First posted 2003-01-27 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2003-08

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Gliosarcoma | interventions — Carmustine; Ethanol

INTERVENTIONS:
Drug: carmustine in ethanol
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of carmustine in treating patients who have progressive or recurrent glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of intratumoral carmustine in ethanol (DTI-015) in patients with unresectable recurrent glioblastoma multiforme. (Phase I of this study closed to accrual as of 01/15/2002.)
* Determine the qualitative and quantitative toxicity of this regimen in these patients.
* Assess the activity of this regimen in these patients.
* Estimate peripheral blood carmustine levels in these patients treated with this regimen.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive carmustine in ethanol (DTI-015) intratumorally over 5 minutes during stereotactic biopsy or open craniotomy.

Cohorts of 3-6 patients receive escalating doses of DTI-015 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 6 patients experience dose-limiting toxicity. (Phase I of this study closed to accrual as of 01/15/2002.)

Additional patients then receive treatment with DTI-015 at the recommended phase II dose.

Patients are followed at 4, 8, and 12 weeks and then every 1-3 months until disease progression.

PROJECTED ACCRUAL: A total of 12 patients were accrued for phase I of this study and approximately 14-18 patients will be accrued for phase II of this study. (Phase I of this study closed to accrual as of 01/15/2002.)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven supratentorial malignant glioblastoma multiforme

  * Clear evidence of disease progression by MRI
  * Unresectable tumor that has spherical, spheroid, or ovoid shape (not multicentric or multilobulated)
  * Central necrosis and/or central cystic areas allowed in the presence of enhancing rim thickness greater than 5 mm
  * No brainstem (pons or medulla) or midbrain (mesencephalon) involvement
  * No involvement of primary sensorimotor cortex in the dominant hemisphere or within 1.5 cm of the optic chiasm, either optic nerve, or any other cranial nerve
  * No tumor extension into the ventricular system
  * Tumor volume no greater than 33.4 cm3
* At least one prior radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No evidence of bleeding diathesis

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* SGOT/SGPT no greater than 2.5 times normal

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 40 mL/min
* BUN no greater than 30 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active uncontrolled infection
* Afebrile unless fever due to presence of tumor
* No other concurrent serious medical or psychiatric illness that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin including Gliadel wafer therapy) and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* No prior intracranial brachytherapy

Surgery:

* Recovered from any prior surgery

Other:

* No prior anticoagulants
* No other concurrent investigational agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Gene David Resnick, MD, Study Chair — Millennix
Locations (12):
- United States (12):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Cancer Center, Denver, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Evanston Northwestern Health Care, Evanston, Illinois
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Barrett Cancer Center, Cincinnati, Ohio
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Massey Cancer Center, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin